CLINICAL TRIAL: NCT01184469
Title: Prospective Observational Study of Peri-implantation Serum hCG Levels
Status: Completed | Type: Observational
Sponsor: Bruce Shapiro M.D. (Industry)
Responsible Party: Sponsor-Investigator, Bruce Shapiro M.D., Medica Director, Fertility Center of Las Vegas
Organization: Fertility Center of Las Vegas (Industry)
Other Study IDs: SAIRB 10-0007
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fresh embryo transfers: Patients who received fresh blastocyst transfer
- Thawed embryo transfers: Patients who received transfers of frozen/thawed embryos

SUMMARY:
The purpose of this study is to prospectively define a set of data suitable for developing models of pregnancy viability. Those models will be based on serum hCG concentration measured during the peri-implantation period in patients that received fresh embryo transfer and those that received transfer of frozen-thawed embryos, and to compare and contrast these models. This may reveal insights into differences between these types of IVF cycles.

DETAILED DESCRIPTION:
The current study seeks to examine the effect of the timing of implantation (as indicated by the first increase in serum hCG level) on the viability of pregnancies and to determine if such effect of timing differs between fresh embryo transfers and frozen-thawed embryos transfers. In this case, the timing of implantation will be measured through serum hCG analysis on days 3, 4, 5, and 7 after blastocyst transfer.

ELIGIBILITY:
Inclusion Criteria:

* IVF patients (adults) who received blastocyst transfer

Exclusion Criteria:

* Those patients using different laboratories

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IVF patients
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy | 10 weeks gestation
  Fetal heart motion at 10 weeks gestation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Center of Las Vegas, Las Vegas, Nevada, United States